CLINICAL TRIAL: NCT04090372
Title: Digital Preop-planning of Total Hip Arthroplasties in Orthopedic
Brief Title: Digital Preop-planning of Total Hip Arthroplasties
Acronym: PLANORTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14 7426 15
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Orthopedic Disorder
Keywords: Osteoarthritis; Hip; Total hip arthroplasty; leg discrepancy; preoperative planning
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group will be assessed by standard preop planning using implants templates.
  Interventions: Device: evaluation of pre-op planning using Traumacad
- TraumaCad Group (Active Comparator): TraumaCad Group will be assessed by preop planning using Traumacad
  Interventions: Device: evaluation of pre-op planning using Traumacad

INTERVENTIONS:
Device: evaluation of pre-op planning using Traumacad — The study will be compare pre-op planning with standard condition or with TraumaCad

SUMMARY:
Residual leg length discrepancy is a common issue after total hip arthroplasty(THA). Digital preoperative planning may improve the accuracy of the surgical procedure and may help the surgeon to precisely predict implants sizes

DETAILED DESCRIPTION:
Total hip arthroplasties (THAs) are used to restore locomotion. More than 150,000 THAs are performed each year in France. Better outcomes require a restoration of limb lengths and anatomy. Post-operative discrepancy is the main cause of complaints and financial compensation in the US after THA. As such, the investigators aim to use preoperative digital planning using TraumaCad to optimize the restoration of the center of rotation of the hips. Preoperative planning are usually performed using anteroposterior standard radiographs, which are scaled to an inaccurate scale. The TraumaCad system (Brainlab®) allows the adjustment of the scales to each patient and the virtual positioning of the implants in order to simulate the intervention for the restitution of the geometrical parameters of the hip.

ELIGIBILITY:
Inclusion Criteria:

* being older than18 years,
* osteoarthritis as the indication for THA

Exclusion Criteria:

* THAs after femoral neck fractures,
* revision surgery,
* major architectural anomaly (Bone tumor, prior fracture of the pelvis, hip dysplasia),
* patients under legal protection,
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
postoperative residual discrepancy | day 3
  The primary endpoint is the postoperative residual discrepancy measured on the radiographs on postop day 3 in millimeter compared using standard planning methods compared to TraumaCad.

SECONDARY OUTCOMES:
comparisons of the reproducibility of the femoral implants sizes | day 3
  Secondary endpoints is comparisons of the reproducibility of the femoral implants sizes predicted by the software
comparison of pelvis parameters | day 3
  Secondary endpoints is the comparison of pelvis parameters in the 2 groups (offset, positioning of the implants) postoperatively. The angle of femur axis and the center of rotation of hip will be measure on the radiography of day 3

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Reina, MD, Principal Investigator — CHU de Toulouse, France
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No